CLINICAL TRIAL: NCT04525742
Title: COVID-19 Pandemic From the Perspective of Parents of Disabled Children
Brief Title: COVID-19 Pandemic and Parents of Disabled Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Berrin Hüner, Medical Doctor, Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 105
Record Dates: First submitted 2020-06-28; First posted 2020-08-25 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: COVID-19; Disabilities Multiple; Cerebral Palsy; Muscular Dystrophies
Keywords: cerebral palsy; COVID-19; pandemic; disability
MeSH Terms: conditions — COVID-19; Cerebral Palsy; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: One study group will be researched- only disabled children's parents, in one arm -way
Masking Description: No masking will be done
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parents who have a disabled child or children (Other): Parents having disabled child or children will be included in the research and it will be wanted to complete the survey questionary
  Interventions: Other: Difficulties lived by disabled children's parents in the period of COVID-19 pandemic

INTERVENTIONS:
Other: Difficulties lived by disabled children's parents in the period of COVID-19 pandemic — It will be a cross sectional study to obtain the information on difficulties lived by disabled children's parents during recent pandemic period

SUMMARY:
Pandemic period could affect the disabled children's rehabilitation and follow-up negatively because of preventive measures and this could create adverse results on their parents.

In this research, it is aimed to determine the positive and negative effects of pandemic on parents and disabled children and to provide an insight for future solutions.

DETAILED DESCRIPTION:
To determine the effect of COVID-19 pandemic and the possible difficulties experienced by the parents of disabled children, a questionnaire was prepared. It takes approximately 10-15 minutes to complete the survey. Questionnaire is loaded to qualtrics program and sent to the families by e-mail or social media accounts.

ELIGIBILITY:
Inclusion Criteria:

* Having disabled child/children
* Having ability and facility to use internet
* Having ability to read and write
* Having enough cognitive capacity to answer the questionnaire
* To accept to participate the research

Exclusion Criteria:

* Not having disabled child/children
* Not having ability and facility to use internet
* Not having ability to read and write
* Not having enough cognitive capacity to answer the questionnaire
* Not to accept to participate the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
A questionnaire that we created will be used to determine the difficulties experienced by disabled children's parents during Covid 19 pandemic related to their medical follow-up | 4 weeks
  Difficulties related to rehabilitation facilities, other medical conditions or ortosis could increase because of Covid 19 pandemic unique conditions

SECONDARY OUTCOMES:
The Fear of COVID-19 Scale | 4 weeks
  The Fear of COVID-19 Scale, a seven-item scale, has robust psychometric properties. It is reliable and valid in assessing fear of COVID-19 among the general population and will also be useful in allaying COVID-19 fears among individuals. Score is minimum 7 pointts and maximum 35 points.

CONTACTS AND LOCATIONS:
Overall Officials: Resa Aydin, Professor, Principal Investigator — İstanbul University İstanbul Faculty of Medicine; Evrim Karadağ Saygı, Professor, Principal Investigator — Marmara University Faculty of Medicine; Özden Özyemisçi Taşkıran, Professor, Principal Investigator — Koc University Faculty of Medicine; Nalan Çapan, Professor, Principal Investigator — İstanbul University İstanbul Faculty of Medicine; Ebru Yilmaz Yalçınkaya, Professor, Study Director — Health Science University
Locations (1):
- Health Science University Gaziosmanpasa Training and Research Hospital, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol was established by Berrin Huner and Ebru Yilmaz Yalcınkaya Statistical analysis (Power analysis) was established by Ozden Ozyemisci Taskiran Informed consent was written by Berrin Huner
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Research is planned to bu conducted between June 15 th and July 15 th 2020. After 15 th of July in 1 week coming statistical analysis will be finished and than in 3 weeks article will be written
Access Criteria: In necessary cases colleced data from the research will be shared with the local ethical committe

REFERENCES:
- [Background] Ahorsu DK, Lin CY, Imani V, Saffari M, Griffiths MD, Pakpour AH. The Fear of COVID-19 Scale: Development and Initial Validation. Int J Ment Health Addict. 2022;20(3):1537-1545. doi: 10.1007/s11469-020-00270-8. Epub 2020 Mar 27. PMID 32226353